CLINICAL TRIAL: NCT04805099
Title: Real-world Safety and Efficacy Data of Checkpoint Inhibitors in Patients With Cancer and Underlying Autoimmune Disease: the Experience of the Hellenic Cooperative Oncology Group
Brief Title: Checkpoint Inhibitors in Patients With Cancer and Underlying Autoimmune Disease
Acronym: CIAD
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: AutoImmune2021
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Autoimmune Diseases; Checkpoint Inhibitor; Immunotherapy
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Checkpoint inhibitor — Treatment with checkpoint inhibitors in patients with preexisting autoimmune disease

SUMMARY:
Patients with cancer and concurrent autoimmune diseases (AID) have been universally excluded from clinical trials evaluating immunotherapy. Data on the safety and efficacy of checkpoint inhibitors in patients with underlying AID is limited. The investigators performed a retrospective multicenter review of medical records of patients with diverse tumor types and underlying AID who received checkpoint inhibitors at Departments of Oncology, affiliated with the Hellenic Cooperative Oncology Group (HeCOG). The primary endpoint was progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients with cancer
* Patients with autoimmune disease
* Treated at HeCOG-affiliated Departments of Oncology
* Early-stage or metastatic

Exclusion Criteria:

* diagnosis of the autoimmune disease after initiation of immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diverse tumor types (early-stage or metastatic) who had received checkpoint inhibitors at HeCOG-affiliated Departments of Oncology Eligible patients had a history of AID, and had received treatment with checkpoint inhibitors as any of line of treatment
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
progression-free survival | Through the completion of the study, for an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hellenic Oncology Cooperative Group, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fountzilas E, Lampaki S, Koliou GA, Koumarianou A, Levva S, Vagionas A, Christopoulou A, Laloysis A, Psyrri A, Binas I, Mountzios G, Kentepozidis N, Kotsakis A, Saloustros E, Boutis A, Nikolaidi A, Fountzilas G, Georgoulias V, Chrysanthidis M, Kotteas E, Vo H, Tsiatas M, Res E, Linardou H, Daoussis D, Bompolaki I, Andreadou A, Papaxoinis G, Spyratos D, Gogas H, Syrigos KN, Bafaloukos D. Real-world safety and efficacy data of immunotherapy in patients with cancer and autoimmune disease: the experience of the Hellenic Cooperative Oncology Group. Cancer Immunol Immunother. 2022 Feb;71(2):327-337. doi: 10.1007/s00262-021-02985-6. Epub 2021 Jun 23. PMID 34164709